CLINICAL TRIAL: NCT06649916
Title: Autism Word Learning and Infant Directed-Speech
Brief Title: Word Learning From Parentese in Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Dr. Pumpki Lei Su, Assistant Professor, The University of Texas at Dallas
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-24-616; R21DC021803 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Autism; Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: autism; word learning; language development
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parentese (Experimental): All participants will learn novel words in two conditions (parentese vs adult register) in each of the experiment (video and live word learning). In the Parentese condition, participants will listen to sentences that contain novel words in parentese.
  Interventions: Behavioral: Parentese Speech
- Adult Register (Active Comparator): All participants will learn novel words in two conditions (parentese vs adult register) in each of the experiment (video and live word learning). In the Adult Register condition, participants will listen to sentences that contain novel words in adult register speech.
  Interventions: Behavioral: Adult Registered Speech

INTERVENTIONS:
Behavioral: Parentese Speech — Novel words are introduced in parentese, a type of speech that is typically characterized by greater pitch variation, longer duration, and louder volume
  Other Names: Infant-Directed Speech
  Arms: Parentese
Behavioral: Adult Registered Speech — Novel words are introduced in standard adult register.
  Other Names: Adult-Directed Speech
  Arms: Adult Register

SUMMARY:
The overall objective of this research is to determine whether parentese delivered in the video format (Aim 1) and in live interaction (Aim 2) facilitates novel word learning in autistic children and to investigate if there are factors that influence the effect of parentese on word learning (Aim 3).

DETAILED DESCRIPTION:
Caregivers frequently use parentese, also known as infant-directed speech (IDS), when speaking to young children. Compared to adult registered speech, parentese is typically characterized by greater pitch variation, longer duration, and louder volume. Parentese facilitates early language development in typically developing (TD) children. However, it remains unknown whether the facilitative effect of parentese on language learning can be generalized to clinical populations such as autistic children given that core autism features (e.g., sensory and social communication differences) may interact with how they process and learn from parentese. Most autistic children do not reach age-appropriate language ability even if they receive timely early intervention. Determining if autistic children can learn language from parentese, a common way language input is provided to young children, is a critical first step toward understanding whether language input needs to be adjusted to optimize their language development.

The overall objective of this research is to determine whether parentese facilitates novel word learning in autistic children and to investigate if the effect of parentese is conditional upon input factors (recorded parentese vs live parentese presented in social interaction) and child factors (extreme responses to auditory input, social motivation). In Aim 1, the investigators will use a video-based word learning paradigm to determine the effect of recorded parentese on novel word learning in autistic children compared to language-matched TD peers. Aim 2 focuses on the effect of live parentese on novel word learning: an experimenter will teach children two novel words, presented in live parentese or live parentese, during social interaction. Aim 3 will examine whether child factors (extreme responses to auditory input, social motivation) explain variability in word learning accuracy from recorded parentese and live parentese in the autistic group. Children's extreme responses to auditory input (including hyper- and hypo-responsiveness) and social motivation will be measured using caregiver questionnaires and will be used to predict word learning accuracy from recorded parentese (Aim 1) and live parentese (Aim 2) in the autistic group.

ELIGIBILITY:
Inclusion Criteria:

* children with or without a diagnosis of ASD between 18 and 59 months

Exclusion Criteria:

* hears another language more than 10% of time based on parent report
* has uncorrected visual impairment or hearing impairment
* has developmental disorders or medical conditions other than ASD that affect language or cognition (excepting psychiatric conditions often comorbid with ASD such as ADHD)

Ages: 18 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of time during which children's eye gaze is directed toward the target object | 300 ms after the target words are introduced
  Children's eye gaze is recorded as they look at images. The proportion of time during which gaze is directed to an image of the targeted word is the dependent measure.

CONTACTS AND LOCATIONS:
Overall Officials: Pumpki L. Su, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This was what was proposed in the study dissemination plan: Summary results of the primary outcomes for all aims will be uploaded to ClinicalTrials.gov within 12 months of the data collection for the final participants.